CLINICAL TRIAL: NCT03947515
Title: Urinary and Prostate Microbiotes and Prostate Cancer
Acronym: MICROPROSTK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-API-02
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cancer group (Experimental)
  Interventions: Procedure: prostate biopsy; Other: Urinary sampling; Other: Rectal swabbing before biopsies are performed
- control group (Experimental)
  Interventions: Procedure: prostate biopsy; Other: Urinary sampling; Other: Rectal swabbing before biopsies are performed

INTERVENTIONS:
Procedure: prostate biopsy — All patients included, will report to the urology department on the date previously agreed with the surgeon. The patient will be seen by the nurse and urologist on duty as part of outpatient care or, more rarely, in ambulatory care. After verification of the patient's identity, the signature of informed consent, the absence of immediate contraindications to biopsy (haemorrhagic and infectious) and the patient's proper preparation (antibiotic prophylaxis and possible enema), the patient will be installed for the taking of samples covered by the protocol (rectal swabbing and prostate biopsies, see paragraph IX). If the patient has not taken the antibiotic prophylaxis or performed the enema, he or she will be reconvened at a later date for the biopsies. After the prostatic biopsies have been performed, the patient's participation in the study ends and his follow-up resumes according to the recommendations adapted to his pathology.
Other: Urinary sampling — It will be collected after the prostate massage performed by the surgeon in charge of the patient during his clinical examination for prostate cancer screening. After elimination of the first draft, the urine will be collected in 2 tubes with borated preservative
Other: Rectal swabbing before biopsies are performed — A rectal swab will then be taken by the urologist on the day the prostate biopsies are taken. The analysis of the digestive microbiota will eliminate contamination of prostate biopsies by bacteria from the faecal flora during transrectal sampling

SUMMARY:
In recent decades, the cancer process has been linked to microbial infections, particularly in gastric and Helicobacter pylori cancers, but also in cervical cancers promoted by exposure to Human papilloma virus (HPV). More recently, it has been shown that bacteria in the intestinal microbiota could promote the development of colorectal cancer by modulating the inflammatory response within the intestinal mucosa. Among male cancers, prostate cancer is the leading cause in France with 54,000 new cases per year. In addition, the dogma that urine is sterile has been broken and the notion of the presence of a "urinary microbiota" in asymptomatic patients is now accepted.

While the risk factors associated with this cancer have not yet been clearly elucidated, recent evidence in the literature agrees that chronic inflammation associated with prostate infection plays a key role as a factor that may promote the development and/or progression of prostate cancer. Most recently, a study shows for the first time that a group of 6 bacteria is found significantly higher in the urine of patients with prostate cancer than in patients with prostate adenoma. Interestingly, clinical microbiology studies conducted at the bacteriology laboratory of the University Hospital of Nice on A. schaalii have shown that this species is also isolated in the urine of patients with bladder and prostate cancers.

The investigators wish to study the association of the 6 bacterial species mentioned above with prostate cancer by directly analyzing the prostate tissue of patients with this condition.

the staff will carry out a multicenter case-control study by recruiting a total of 260 patients in 4 centres (Nice coordinating centre, Marseille, Tours and Nîmes): 130 in the prostate cancer group and 130 in the prostate adenoma control group. This project is a research involving the human person of category 2.

The innovative aspect of the work consists in detecting and quantifying in situ in the prostate tissue the presence of these 6 bacterial species per culture and per PCR in real time, comparing the prostate microbiota in terms of richness and diversity between cancer patients and those without cancer. Ultimately, this study opens up exciting prospects with the possibility of determining a microbial origin of prostate cancer and considering antibiotic therapy for anti-cancer purposes such as H. pylori and gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* Male sex
* Patient with a prostate biopsy programmed for suspected prostate adenocarcinoma on elevation of PSA and/or TR suspect and/or MRI suspect
* Signed Informed Consent
* Affiliation to a social security system

Exclusion Criteria:

* Taking systemic antibiotic treatment (per os or I.V.) within 3 months before inclusion.
* Contraindications to the performance of an ultrasound-guided transrectal prostate biopsy: coagulation disorders and urogenital infections.
* History of surgical treatment of the urinary and genital tract within 6 months before inclusion
* Person under guardianship, curatorship or unable to express consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Number of 6 bacterial species in prostate biopsy | 48 months
  detection in prostate biopsy by real-time PCR and/or culture followed by identification by MALDI-TOF mass spectrometry of at least one of the following 6 bacterial species : S. anginosus, V. cambriense, P. lymphophilum, A. lactolyticus, A. obesiensis and A. schaalii.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Cannes hospital, Cannes
  - marseille Hospital, Marseille
  - nice Hospital, Nice
  - Tours hospital, Tours

IPD SHARING:
Plan to Share IPD: No